CLINICAL TRIAL: NCT05416814
Title: Safety and Feasibility of Kefir Administration in Critically Ill Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lioudmila Karnatovskaia, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-005687
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness | interventions — Kefir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kefir administration in critically ill adults (Experimental): Critically ill subjects will receive Kefir throughout the length of their ICU course in an ascending dosing regimen
  Interventions: Dietary Supplement: Kefir

INTERVENTIONS:
Dietary Supplement: Kefir — Oral route (via feeding tube in intubated patients). Serving size 240mL to be given in an ascending dosing regimen if tolerated starting at 60 mL/day, 120 mL/day until single 240 mL/day; if evidence of intolerance, dose will be reduced to previously tolerated dose.
  Other Names: Lifeway Foods® Original Kefir Unsweetened Whole Milk

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of kefir administration in critically ill adults.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult patients receiving antibiotics.
* Functional GI tract (able to tolerate oral diet or tube feeding).

Exclusion Criteria:

* Received antibiotics for >72 hours prior to enrollment.
* Known immunosuppression (due to medications including chronic steroids, TNF-alpha inhibitors, monoclonal antibodies, immunosuppressive antimetabolites, etc.).
* Compromised gut integrity (bowel resection, GI malignancy, GI bleed, inflammatory bowel disease).
* History of CDI within 60 days.
* Liver failure or pancreatitis.
* Dairy intolerance or milk allergy.
* Patients consuming probiotics at baseline.
* Artificial heart valve.
* Extremely poor prognosis and not expected to survive the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Number of adverse effects related to kefir administration including vomiting, aspiration, diarrhea, interactions with medications or tube feeds, bacteremia secondary to a bacterium in kefir
Feasibility of Kefir administration | 30 days
  Number of subjects to have more than 75% of doses given when subject is allowed to have PO/feeding tube administration and are tolerated

CONTACTS AND LOCATIONS:
Overall Officials: Lioudmila Karnatovskaia, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta VK, Rajendraprasad S, Ozkan M, Ramachandran D, Ahmad S, Bakken JS, Laudanski K, Gajic O, Bauer B, Zec S, Freeman DW, Khanna S, Shah A, Skalski JH, Sung J, Karnatovskaia LV. Safety, feasibility, and impact on the gut microbiome of kefir administration in critically ill adults. BMC Med. 2024 Feb 20;22(1):80. doi: 10.1186/s12916-024-03299-x. PMID 38378568
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials